CLINICAL TRIAL: NCT05987696
Title: Phase I Study to Evaluate the Safety and Efficacy of NK Cell Therapy in Acute Myeloid Leukemia (AML).
Brief Title: Natural Killer(NK) Cell Therapy in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hangzhou Qihan Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023028
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: AML, Adult; Minimal Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Cyclophosphamide; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CD33/CLL1 dual CAR-NK cell (Experimental): CLL1/CD33 dual CAR-NK cell therapy in Adult subjects with r/r AML
  Interventions: Drug: CD33/CLL1 dual CAR-NK cell; Drug: Cyclophosphamid; Drug: Fludarabine; Drug: Cytarabine
- CD33 CAR-NK cell (Experimental): CD33 CAR-NK cell therapy in Adult subjects with r/r AML
  Interventions: Drug: Cyclophosphamid; Drug: Fludarabine; Drug: Cytarabine; Drug: CD33 CAR-NK cell
- super NK cell (Experimental): super NK cell therapy in Adult subjects with AML MRD
  Interventions: Drug: Cyclophosphamid; Drug: Fludarabine; Drug: Cytarabine; Drug: super NK cell

INTERVENTIONS:
Drug: CD33/CLL1 dual CAR-NK cell — NK cell therapy
  Arms: CD33/CLL1 dual CAR-NK cell
Drug: Cyclophosphamid — Lympho-conditioning Agent
Drug: Fludarabine — Lympho-conditioning Agent
Drug: Cytarabine — Lympho-conditioning Agent
Drug: CD33 CAR-NK cell — NK cell therapy
  Arms: CD33 CAR-NK cell
Drug: super NK cell — NK cell therapy
  Arms: super NK cell

SUMMARY:
This is a phase 1, first-in-human (FIH), open-label, multicohort study to evaluate the safety, tolerability and preliminary efficacy of iPSC NK cells in patients with relapsed/refractory AML or AML Minimal Residual Disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF).
2. ≥18 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 and life expectancy greater than 12 weeks.
4. Diagnosis of r/r AML (Cohort 1 and 2) or AML MRD (Cohort 3).
5. Cohort 1: Both CLL1 and CD33 expression are positive in AML blasts; Cohort 2: The expression of CD33 in AML blast is positive.
6. Adequate organ and marrow function, as defined below:

   1. Blood creatinine (Cr) ≤ 2 x ULN or calculated creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min;
   2. Total bilirubin (TBIL) ≤ 2 x the ULN;
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN;
   4. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN;
7. Females of childbearing potential must have a negative serum pregnancy test.
8. Donor specific antibody (DSA) is negative: MFI <= 2000.

Exclusion Criteria:

1. Allergic to drug used in this study.
2. Subjects received any antitumor therapy as follows, prior to first NK infusion:

   1. Systemic steroid therapy within 3 days (except physiological replacement therapy);
   2. Systemic antitumor therapy within 2 weeks or at least 5 half-lives, whichever is less;
   3. Radiotherapy within 4 weeks;
   4. Donor lymphocyte infusion within 6 weeks;
   5. Intrathecal treatment within 1 week;
   6. CAR-T therapy, CAR-NK therapy, or any other genetically modified cell therapy product within 6 months;
3. History of allogeneic stem cell transplantation.
4. Received the vaccine within 4 weeks prior to the first infusion and/or expected to require vaccination from the study period to 12 weeks after the last infusion.
5. Active central nervous system Leukemia.
6. Acute Promyelocytic Leukemia (APL).
7. History of other malignant tumors, except for those who have achieved complete remission more than 5 years after radical treatment without any signs of recurrence.
8. Active autoimmune diseases.
9. History of central nervous system disease or meningeal involvement such as epilepsy, paralysis, aphasia, stroke, etc.
10. Serious cardiovascular and cerebrovascular diseases:

    1. Severe heart rhythm or conduction abnormalities, corrected QT interval (QTc)≥480 ms;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events within 6 months prior to first infusion;
    3. New York Heart Association (NYHA) class II or above congestive heart failure or left ventricular ejection fraction (LVEF) <50% in color Doppler echocardiography;
    4. Hypertension that cannot be controlled by drug.
11. Active pulmonary infection; SpO2 ≤90%; Pulmonary embolism, chronic obstructive pulmonary disease, or interstitial lung disease.
12. Uncontrolled bacterial, fungal, or viral infection. Known HIV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection.
13. History of substance abuse.
14. Toxicity induced by previous therapy not recovered to ≤ grade 2(NCI-CTCAE v5.0).
15. Large surgical treatment within 4 weeks prior to first infusion, not including diagnostic biopsy.
16. Pregnant/breastfeeding women.
17. Investigator-assessed presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 Days from first dose of iPSC NK cell infusion
Incidence of subjects with Dose Limiting Toxicities within each dose level cohort | 28 Days from first dose of iPSC NK cell infusion

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | Up to approximately 2 years after last dose of iPSC NK cell infusion
MRD negative rate | 28 Days from first dose of iPSC NK cell infusion
Event-free survival | Up to approximately 2 years after last dose of iPSC NK cell infusion]
Relapse-free survival | Up to approximately 2 years after last dose of iPSC NK cell infusion
Overall survival (OS) | Up to approximately 2 years after last dose of iPSC NK cell infusion
Determination of the pharmacokinetics (PK) of iPSC NK cells in peripheral blood | Up to approximately 2 years after last dose of iPSC NK cell infusion
  The PK of iPSC NK in peripheral blood will be reported as the relative percentage of product DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China